CLINICAL TRIAL: NCT00340548
Title: Host Genetic Factors Influencing HIV1 and HCV Viral Loads and AIDS Clinical Progression in a Hemophilia Cohort (HGDS-3)
Status: Terminated | Type: Observational
Why Stopped: lapse in IRB review
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902173; 02-C-N173
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Hemophilia; AIDS
Keywords: Genotyping; Polymorphisms; Co-Infection; Chemokines; Associations; HIV; HCV; Hepatitis C; Hemophilia
MeSH Terms: conditions — Hemophilia A; Acquired Immunodeficiency Syndrome; Coinfection; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

Over 80% of the hemophiliac population who became infected with HIV prior to 1985 are also co-infected with HCV. Thus, hemophiliacs represent an important population for studies of the natural history of these chronic viral infections.

Moreover, the high rate of co-infection makes it an ideal group for assessing the interaction between the viruses and the relationship between viral specific immune responses and clinical progression.

Although the hemophiliac poulation is unique, co-infection by these chronic viral pathogens is becoming increasingly common, particularly amongst intravenous drug users, who account for approximately 25% of the HIV-1 epidemic in the United States.

Objectives:

The aim of this study is to determine if polymorphism in the promoter region of TH1 and Th2 cytokines are associated with (1) intracellular cytokines levels in CD4 + Tcells, (2) Human Immunodeficiency Virus (HIV) and Hepatitis C virus (HCV) viral loads, and (3) clinical progression of HIV1 to AIDS in hemophiliacs.

Eligibility:

The current proposal will investigate host genetic factors related to HIV-1 and HCV immunopathogenesis by studying children and adolescents enrolled in the Hemophilia Growth and Development Study (HGDS).

Design:

This study is in collaboration with the principle investigators of the Hemophilia Growth and Development Study (HGDS) as part of a grant "Pathogenesis of HIV and HCV in Hemophilia: HGDS-3" with funding support by NIH/NICHD for the period 9/25/01 through 8/31/2005.

This multicenter, United States study represents a well-characterized, prospectively followed cohort of HCV-infected hemophiliacs, of whom 207 are HIV-1 co-infected.

Enrollment of the hemophiliac cohort was completed between 3/89 and 6/90. The final observation of the cohort (follow-up 16) was concluded during 7/98. No new samples or clinical data will be collected on this population.

The LGD plays two roles in this project: (1) an administrative role overseeing the withdrawal, handling, and transport of samples from the HGDS/LGD and central repositories at the NCI-Frederick, and (2) a scientific role continuing investigations to determine the role of host genetic factors in Th1 and Th2 immune response and regulation of HCV and HIV viral replication..

DETAILED DESCRIPTION:
Background:

Over 80% of the hemophiliac population who became infected with HIV prior to 1985 are also co-infected with HCV. Thus, hemophiliacs represent an important population for studies of the natural history of these chronic viral infections.

Moreover, the high rate of co-infection makes it an ideal group for assessing the interaction between the viruses and the relationship between viral specific immune responses and clinical progression.

Although the hemophiliac poulation is unique, co-infection by these chronic viral pathogens is becoming increasingly common, particularly amongst intravenous drug users, who account for approximately 25% of the HIV-1 epidemic in the United States.

Objectives:

The aim of this study is to determine if polymorphism in the promoter region of TH1 and Th2 cytokines are associated with (1) intracellular cytokines levels in CD4 + Tcells, (2) Human Immunodeficiency Virus (HIV) and Hepatitis C virus (HCV) viral loads, and (3) clinical progression of HIV1 to AIDS in hemophiliacs.

Eligibility:

The current proposal will investigate host genetic factors related to HIV-1 and HCV immunopathogenesis by studying children and adolescents enrolled in the Hemophilia Growth and Development Study (HGDS).

Design:

This study is in collaboration with the principle investigators of the Hemophilia Growth and Development Study (HGDS) as part of a grant "Pathogenesis of HIV and HCV in Hemophilia: HGDS-3" with funding support by NIH/NICHD for the period 9/25/01 through 8/31/2005.

This multicenter, United States study represents a well-characterized, prospectively followed cohort of HCV-infected hemophiliacs, of whom 207 are HIV-1 co-infected.

Enrollment of the hemophiliac cohort was completed between 3/89 and 6/90. The final observation of the cohort (follow-up 16) was concluded during 7/98. No new samples or clinical data will be collected on this population.

The LGD plays two roles in this project: (1) an administrative role overseeing the withdrawal, handling, and transport of samples from the HGDS/LGD and central repositories at the NCI-Frederick, and (2) a scientific role continuing investigations to determine the role of host genetic factors in Th1 and Th2 immune response and regulation of HCV and HIV viral replication..

ELIGIBILITY:
* INCLUSION CRITERIA:

The current Study will involve analysis of existing samples (DNA, serum, cells, plasma) and data. The entire set of 333 subjects in the HGDS cohort will be analyzed.

EXCLUSION CRITERIA:

No subjects will be excluded from the HGDS cohort.

Ages: 4 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2002-04-09; Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

PRIMARY OUTCOMES:
Receipt of 333 samples | Annually

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W McVicar, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (15):
- United States (15):
  - University of California, San Diego, La Jolla, California
  - Childrens Hospital, Los Angeles, Los Angeles, California
  - St. Vincent Hospital & Health Care Center, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Tulane University, New Orleans, Louisiana
  - NCI Frederick Cancer Research Center, Frederick, Maryland
  - Wayne State University Hutzel Hospital, Detroit, Michigan
  - Childrens Mercy Hospital, Kansas City, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Cornell University, New York, New York
  - Mt. Sinai Medical Center, New York, New York
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Milton Hershey Medical Center, Hershey, Pennsylvania
  - University of Texas, Houston, Houston, Texas
  - University of Texas, San Antonio, San Antonio, Texas

REFERENCES:
- [Background] Dean M, Carrington M, Winkler C, Huttley GA, Smith MW, Allikmets R, Goedert JJ, Buchbinder SP, Vittinghoff E, Gomperts E, Donfield S, Vlahov D, Kaslow R, Saah A, Rinaldo C, Detels R, O'Brien SJ. Genetic restriction of HIV-1 infection and progression to AIDS by a deletion allele of the CKR5 structural gene. Hemophilia Growth and Development Study, Multicenter AIDS Cohort Study, Multicenter Hemophilia Cohort Study, San Francisco City Cohort, ALIVE Study. Science. 1996 Sep 27;273(5283):1856-62. doi: 10.1126/science.273.5283.1856. PMID 8791590
- [Background] Daar ES, Lynn H, Donfield S, Gomperts E, Hilgartner MW, Hoots WK, Chernoff D, Arkin S, Wong WY, Winkler CA; Hemophilia Growth and Development Study. Relation between HIV-1 and hepatitis C viral load in patients with hemophilia. J Acquir Immune Defic Syndr. 2001 Apr 15;26(5):466-72. doi: 10.1097/00126334-200104150-00011. PMID 11391167
- [Background] Daar ES, Lynn H, Donfield S, Gomperts E, O'Brien SJ, Hilgartner MW, Hoots WK, Chernoff D, Arkin S, Wong WY, Winkler CA; Hemophilia Growth and Development Study. Hepatitis C virus load is associated with human immunodeficiency virus type 1 disease progression in hemophiliacs. J Infect Dis. 2001 Feb 15;183(4):589-95. doi: 10.1086/318539. Epub 2001 Jan 12. PMID 11170984
- [Background] Hilgartner MW, Donfield SM, Willoughby A, Contant CF Jr, Evatt BL, Gomperts ED, Hoots WK, Jason J, Loveland KA, McKinlay SM, et al. Hemophilia growth and development study. Design, methods, and entry data. Am J Pediatr Hematol Oncol. 1993 May;15(2):208-18. doi: 10.1097/00043426-199305000-00009. PMID 8498644